CLINICAL TRIAL: NCT06510985
Title: Transcutaneous Vagus Nerve Stimulation (tVNS) for Improved Recovery After Exertion in Patients With Long/Post-COVID.
Brief Title: Transcutaneous Vagus Nerve Stimulation (tVNS) for Improved Recovery After Exertion.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TUE012_tvns_longCovid
Record Dates: First submitted 2024-07-17; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-04

CONDITIONS: Post-COVID-19 Syndrome
Keywords: Post-COVID-19 Syndrome; taVNS; effort; fatigue; heart rate
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring with high/low-intensity stimulation (Experimental): The cross-over design includes one group which starts with high-intensity stimulation (n = 40) and another group, who starts with low-intensity stimulation (n = 40). The first group receives at first high-intensity for 6 weeks, followed by a low-intensity stimulation phase for 6 weeks. To control for placebo effects, other forty individuals start with the 6-week low-intensity stimulation phase followed by 6 weeks of high-intensity tVNS stimulation phase.
  Interventions: Device: transcutaneous vagus nerve stimulation; Behavioral: Monitoring; Device: cardiowatch bracelet
- Monitoring without stimulation (Experimental): Another group of patients is included as a control group (n = 40) undergoing 'treatment as usual' for Long/Post Covid. This group of participants receive the same monitoring throughout their participation during 12 weeks as the Stimulation-Group. As there is no standardized treatment protocol for Long/Post Covid, 'treatment as usual' implies a supportive approach.
  This group of participants have the option to receive taVNS stimulation after participating in the study.
  Interventions: Behavioral: Monitoring; Device: cardiowatch bracelet

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — The study employs a CE-certified tVNS® E device, ensuring European safety standards (EU regulation 2017/745 on medical devices). This device features a stimulation cycle of 28 seconds on and 32 seconds off, with a 25 Hz impulse frequency. For the high-intensity group, the stimulation intensity will be individually adjusted in the session before starting the high-intensity tVNS stimulation at home. Recommended daily usage is max. 4 hours, after which it automatically shuts off.
  Arms: Monitoring with high/low-intensity stimulation
Behavioral: Monitoring — Participants are monitored over 12 weeks using a combination of questionnaires and ecological momentary assessment. This approach allows for a comprehensive assessment of the patient's health and well-being.
Device: cardiowatch bracelet — The study employs the medically certified cardiowatch bracelet from Corsano (CE-MDR medical certification, FDA 510 (k) cleared) for continuous monitoring of vital signals, such as heart rate, heart rate variability, breathing rate, SpO2, physical activity and sleep.

SUMMARY:
Widespread infection with SARS-CoV-2 has resulted in millions of people having Post-COVID. Post-COVID is a complex, non-monolithic disease with diverse clinical manifestations. Symptoms range from fatigue, brain fog, muscle aches and shortness of breath, affecting multiple organ systems simultaneously. To directly address this multi-organ component of Post-COVID, innovative treatment methods are urgently needed. One potential treatment that we will investigate in our study, is the intervention via the vagus nerve, as the cranial nerve plays a central role in communication between the body and the brain and influences targeted behavior. This innovative approach is based on our clinically relevant findings regarding the effects where acute tVNS increased the level of effort (Neuser et al., 2020; Ferstl et al., 2021), specifically targeting a key symptom of Post-COVID. In the proposed study, the investigators aim to investigate the effectiveness of transcutaneous vagus nerve stimulation (tVNS) as a non-invasive, self-administered treatment for Post-COVID symptoms at home. To evaluate the clinically relevant effects of repeated taVNS application (high-intensity stimulation), the investigators will employ a randomized cross-over design to investigate stimulation-induced changes in fatigue, depression and motivation to work for reward compared to low-intensity stimulation and to a control group.

DETAILED DESCRIPTION:
The proposed study aims to advance the understanding of Post-COVID treatment using a randomized cross-over design to evaluate the taVNS-induced changes over 12 weeks. A hundred twenty patients diagnosed with Long/Post-COVID are randomly assigned to one of three groups related to the two arms of the study ("Monitoring with low/high-intensity stimulation" vs. Monitoring without stimulation"). In the treatment group, forty patients will start with high-intensity taVNS for 6 weeks, then switch to low-intensity stimulation for an additional 6 weeks. Another 40 patients begin with low-intensity stimulation for 6 weeks, followed by high-intensity taVNS stimulation. The control group ("Monitoring without stimulation") is able to receive taVNS after participation in the study.

The treatment group and the control group will participate in the same monitoring procedures. All participants will attend an initial laboratory session to complete several baseline assessments, including questionnaires, measuring energy expenditure via indirect calorimetry and completing a body silhouette task. Blood samples are taken at every session to evaluate changes in metabolic and inflammatory markers. To assess the motivation to work for rewards, the investigators employ an effort-based-cost-benefit paradigm (Effort Allocation Task). All these lab assessments will be repeated after 6 and 12 weeks to evaluate stimulation-induces changes in primary and secondary outcomes. In addition, all participants are given a cardio bracelet to monitor physiological parameters (e.g. heart rate, heart rate variability, breathing, skin conductance, step counts) over the study period. Over the 12 weeks, the treatment group will self-administer taVNS for four hours daily in a targeted manner, anticipating forthcoming exertion and stimulating in anticipation of an effortful event to enhance the patients' motivational drive and recovery. Another essential part of the study is the monitoring over the 12 weeks. All participants will complete daily ecological momentary assessments via smartphone to monitor their mental states. In addition, participants will perform once a day one of two discounting games (effort or temporal discounting task) to investigate changes in their decision behavior over time. The effort discounting task is essential to assess the motivation of post-COVID patients to pursue subjectively effortful situations over the 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* individuals who have previously tested positive for SARS-CoV-2 infection (preferred PCR-Test) or have a medically confirmed history of COVID-19 (preferred SARS-CoV-2 Antibody-test) and have persistent symptoms (including Post-COVID) .
* clinical diagnoses made by physician: individuals are included with at least one persistent symptom for at least 4 weeks (Long-COVID) or at least 8 weeks (Post-COVID) following the SARS-CoV-2 infections, such as fatigue, shortness of breath, brain fog, headaches, irritability, cognitive difficulties, muscle or joint pain, sleep disturbances, etc.
* Participants should not have an alternative explanation for their persistent symptoms, ruling out other medical or psychiatric conditions.

Exclusion Criteria:

* lack of capacity for consent
* insufficient German language skills: Participants must have sufficient (B2 German) language skills to understand the informed consent form, study procedures, and questionnaires.
* Intensive Care Unit treatment during COVID-19 infection
* BMI > 18.5 & BMI < 35 kg/m2

Lifetime (according to DSM 5):

* brain injury, stroke, epilepsy, or history of seizures
* schizophrenia
* bipolar disorder
* severe substance use disorders, except tobacco
* cardiac arrhythmia, coronary heart disease
* 12-month prevalence: pregnancy or nursing

Additional exclusion criteria for a safe application of tVNS:

* active implant (pacemaker, cochlear implant, implanted electrode device) and cerebral shunts
* required permanent use of left-sided hearing aid
* ear infections, open wounds, or impaired skin at electrode sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-19 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Stimulation-induced changes in invigoration: frequency of button presses during the first seconds of the trial to gain monetary rewards in the Effort Allocation Task. | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in invigoration to work for rewards are operationalized as the relative increase in the frequency of button presses on an Xbox controller during the first seconds of the trial in the Effort Allocation Task.
Stimulation-induced changes in symptoms of depression | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in symptoms of depression are measured via the Montgomery Asberg Depression Scale. The MADRS comprises 10 items rated on a scale from 0 to 6 to compute a sum score with higher scores indicating severe symptoms of depression.
Stimulation-induced changes in physical and mental aspects of fatigue | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in fatigue are measured by the Chalder Fatigue scale. The CFS comprises 11 questions rated on a 4-point Likert scale to compute a sum score.
  It will be measured three times six weeks apart.

SECONDARY OUTCOMES:
Stimulation-induced changes in heart rate variability | during 6-week tVNS compared to during 6-week low-intensity stimulation phase
  Changes in heart rate variability are measured by a cardiowatch bracelet to evaluate autonomic nervous system activity.
  It will be measured over three months daily.
Stimulation-induced changes in physical activity | during 6-week tVNS compared to during 6-week low-intensity stimulation phase
  Changes in physical activity are measured by step count per day, which are recorded by the cardiowatch bracelet.
  It will be measured over three months daily.
Stimulation-induced changes in wanting the monetary rewards | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in wanting monetary rewards are measured via a visual analogue scale rating after each effortful trial in the Effort Allocation Task.
  It will be measured three times six weeks apart.
Stimulation-induced changes in exertion | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in exertion are measured via a visual analogue scale rating after each effortful trial.
  It will be measured three times six weeks apart.
Stimulation-induced changes in the motivation to invest effort: the discounting rate reflecting rewards devalued by effort | during 6-week tVNS compared to during 6-week low-intensity stimulation phase
  Changes in the motivation to invest effort is quantified by estimating the participant-specific discounting factor (k) and the inverse temperature parameter (β), which are derived by fitting the participant's observed choice behavior in the effort discounting task to discounting models.
  It will be measured at least twice a week over three months.
Stimulation-induced changes in resting energy expenditure | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in resting energy expenditure are measured by indirect calorimetry. It will be measured three times six weeks apart.
Stimulation-induced changes in metabolic and inflammatory markers | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Metabolic hormone levels and inflammatory markers are assessed from blood samples.
  It will be measured three times six weeks apart.
Stimulation-induced changes in health-related quality of life | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in health-related quality of life are measured by the Short-Form-12 health survey (SF-12), consisting of 12 questions (weighted sum score).
  It will be measured three times six weeks apart.
Stimulation-induced changes in mood | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in positive and negative mood ratings are measured with the PANAS questionnaire (scale 1-5) It will be measured three times six weeks apart.
Stimulation-induced changes in maintenance:the average relative frequency across the complete trial to gain monetary rewards in the Effort Allocation Task. | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Changes in motivation to work for rewards are operationalized as the average relative increase in the frequency of button presses on an Xbox controller across the complete trial in the Effort allocation task.
Stimulation-induced changes in heart rate | during 6-week tVNS compared to during 6-week low-intensity stimulation phase
  Changes in heart rate are measured by a cardiowatch bracelet depending on physical activity phases

OTHER OUTCOMES:
Sensor-based data will be included in exploratory analyses. | during 6-week tVNS compared to during 6-week low-intensity stimulation phase
  Changes in sensory-based data are measured by a cardiowatch bracelet
Changes in Questionnaires | Pre treatment vs. after 6-week tVNS vs. after 6-week low-intensity stimulation phase
  Questionnaires will be included in exploratory analyses and as a confounding variable.

CONTACTS AND LOCATIONS:
Overall Officials: Nils B. Kroemer, Prof. Dr., Principal Investigator — Department of Psychiatry & Psychotherapy, University of Tübingen,Tübingen, 72076; Andreas J. Fallgatter, Prof. Dr., Principal Investigator — Department of Psychiatry & Psychotherapy, University of Tübingen,Tübingen, 72076
Locations (1):
- Department of Psychiatry & Psychotherapy, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany